CLINICAL TRIAL: NCT02202564
Title: Preliminary Results for the Double-dose Adenovirus-mediated Adjuvant Therapy Improving Outcome of Liver Transplantation in Patients With Advanced Hepatocellular Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Huazhong University of Science and Technology (Other)
Collaborators: Beijing YouAn Hospital (Other)
Responsible Party: Principal Investigator, Ding Ma, Director of the Laboratory of Tumor invasion and metastasis, Huazhong University of Science and Technology
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LT-02
Record Dates: First submitted 2014-07-26; First posted 2014-07-29 (Estimated); Last update posted 2014-07-29 (Estimated); Status verified 2014-07

CONDITIONS: Liver Cancer; Hepatocellular Carcinoma
Keywords: hepatocellular carcinoma; liver transplantation; adenovirus-thymidine kinase; gene therapy
MeSH Terms: conditions — Liver Neoplasms; Carcinoma, Hepatocellular | interventions — Liver Transplantation; Ganciclovir

ARMS (2):
- LT+ADV-TK (Experimental): Liver transplantation and double-dose ADV-TK/ganciclovir administration The first ADV-TK dose was administered before closing the peritoneal layer; the second ADV-TK dose was administered 2 months after LT; ganciclovir was slowly administered 36 hours after LT and twice daily for 14 days.
  Interventions: Procedure: LT; Drug: ADV-TK; Drug: ganciclovir
- LT (Active Comparator): Orthotopic liver transplantation
  Interventions: Procedure: LT

INTERVENTIONS:
Procedure: LT — Orthotopic LT
  Other Names: liver transplantation
Drug: ADV-TK
  Other Names: adenovirus-thymidine kinase
  Arms: LT+ADV-TK
Drug: ganciclovir
  Arms: LT+ADV-TK

SUMMARY:
HCC patients with tumors >5 cm in diameter, regardless of involvement in the intrahepatic and extrahepatic portal branches participated in the study. Patients were randomized allocated in liver transplantation (LT) only group and LT plus ADV-TK therapy group. All patients received orthotopic liver transplantation; in the LT plus ADV-TK group, ADV-TK therapy was delivered to patients twice.

ELIGIBILITY:
Inclusion Criteria:

* 18～70 years of age (Male and Female).
* Clinical diagnosis of advanced hepatocellular carcinoma who could accept liver transplantation
* Patients who had unresectable HCC >5 cm and no metastasis in lungs and bones were eligible to participate in this study. Tumor involvement in the intrahepatic and extrahepatic portal branches was not considered to be an exclusion criterion.
* No prior chemotherapy, radiation therapy, targeted therapy or other kind of biological treatment within 4 weeks.
* Provide written informed consent

Exclusion Criteria:

* Metastasis in lungs and bones
* Invasion in main vescular.
* Contraindications of liver transplantation
* Contraindications of operation of other organ system
* Hypersensitivity to adenovirus, GCV or similar drugs
* Accept clinical trials of other drugs
* Immunological deficit
* Active pregnancy
* Unable or unwilling to sign informed consents

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2006-10; Primary Completion 2011-10 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Overall survival rate | up to 3-year
Recurrence-free survival rate | up to 3-year

CONTACTS AND LOCATIONS:
Overall Officials: Ding Ma, M.D., Principal Investigator — Huazhong University of Science and Technology